CLINICAL TRIAL: NCT05225272
Title: Evaluation of the Effectiveness of an Enhanced Recovery After Surgery Protocol in Patients Undergoing On-pump Cardiac Surgery
Brief Title: Effectiveness of an Enhanced Recovery After Surgery Protocol in Patients Undergoing On-pump Cardiac Surgery
Acronym: ERASCs
Status: Not yet recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 21.320
Record Dates: First submitted 2022-01-26; First posted 2022-02-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Disorder; Heart, Functional, Postoperative, Cardiac Surgery
Keywords: On-pump cardiac surgery; Enhanced recovery after surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing on-pump cardiac surgery: The investigators aim to conduct a bidirectional (prospective and retrospective) observational, cohort study including on-pump cardiac surgery patients.
  Interventions: Other: Enhanced Recovery Program for on-pump cardiac surgery

INTERVENTIONS:
Other: Enhanced Recovery Program for on-pump cardiac surgery — Implementation of a Enhanced Recovery Program for on-pump cardiac surgery patients

SUMMARY:
In 2019, the Enhanced Recovery After Surgery (ERAS) Society published recommendations for perioperative care in cardiac surgery. ERAS recommendations included 22 perioperative interventions that may be part of any cardiac Enhanced Recovery Program (ERP). Since that publication, additional perioperative interventions were reported and may be added to a cardiac ERP. Studies on cardiac ERPs report variable benefits on postoperative recovery including lower pain scores, lower opioid consumption and related side effects, shorter intensive care unit and hospital discharge times. At the "Centre Hospitalier de l'Université de Montréal" (CHUM), although most care takers are aware of ERAS recommendations for cardiac surgery patients, adherence to these recommendations is heterogeneous and a cardiac ERP was never implemented.

DETAILED DESCRIPTION:
Primary objective: Estimate the effect of implementation of an ERP (including the use of a checklist and teaching of caretakers) on the time needed for patient extubation after on-pump cardiac surgery.

Secondary objective: Estimate the effect of implementation of a ERP (including the use of a checklist and teaching of caretakers) on the need for reintubation, the need to return to the operating room for hemostasis, on pain scores, opioid consumption and related side effects, on the incidence of postoperative delirium in the intensive care unit, on intensive care unit and hospital discharge times, on postoperative complications (stroke, acute renal failure, postoperative atrial fibrillation), and on in-hospital mortality, 30-day mortality and hospital readmission.

The hypothesis of the study is that implementation of an ERP (including the use of a checklist and teaching of caretakers) in patients undergoing on-pump cardiac surgery improves postoperative recovery through shorter extubation time and a reduction of postoperative complications.

Design of the study: single center, bidirectional (prospective and retrospective) chronological cohort study. The adherence to ERP interventions will be measured.

Prospective data will be collected in eligible patients after implementation of a cardiac ERP and compared retrospectively with eligible patients who had surgery in the year before (but not in the four weeks preceding) implementation of the cardiac ERP. In these patients, prospective data is already collected in a quality of care database in cardiac surgery.

The cardiac ERP will be implemented using a checklist designed by cardiac surgeons, anesthesiologists and intensive care specialists. The checklist is based on official ERAS recommendations and other interventions suggested in further studies on ERAS after cardiac surgery. Professionals involved in the perioperative care of cardiac surgery patients will receive specific ERP teachings three weeks and one week before the official implementation of the cardiac ERP. Posters detailing the cardiac ERP will be clearly visible in the cardiac operating rooms and next to the intensive care unit beds to promote adherence.

ELIGIBILITY:
Inclusion Criteria:

* On-pump cardiac surgery

Exclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) lower than 50%
* Glomerular filtration rate lower than 50 mL/min
* Significant pulmonary hypertension (systolic pulmonary artery pressure higher than 65 mmHg)
* Presence of Intra-aortic balloon pump therapy before surgery
* Endocarditis surgery
* An estimated mortality over 8% based on the EuroSCORE II
* Patients who already had cardiac surgery in the past.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators aim to conduct a bidirectional cohort study including on-pump cardiac surgery patients. This study will take place at the Centre Hospitalier de l'Université de Montréal (CHUM).
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Time before patient extubation | From the end of the surgery to extubation, up to 1 week
  Time elapsed between final wound dressing and removal of the endotracheal tube, before and after implementation of the cardiac ERP.

SECONDARY OUTCOMES:
Incidence of reintubation | Up to 24 hours after extubation
  Need for postoperative endotracheal intubation given the occurrence of respiratory or non-respiratory complication after extubation.
Acute pain scores using the Numerical Rating Scale (NRS) | 8, 16, 24 and 48 hours after surgery
  Using the verbal NRS, where 0 means "no pain" and 10 "worst pain imaginable"
Opioid consumption | 8, 16, 24 and 48 hours after surgery
  Opioid consumption converted in intravenous morphine equivalents
Opioid side effects | 8, 16, 24 and 48 hours after surgery
  Including nausea, vomiting, sedation and pruritus
Incidence of delirium in the intensive care unit (ICU) using the ICDSC score | Up to 7 days after surgery or ICU discharge, whichever comes first
  Delirium will be assessed every 8 hours during the ICU stay using the Intensive Care Delirium Screening Checklist (ICDSC). A total ICDSC score greater or equal to 4 has a 99% sensitivity for a psychiatric diagnosis of delirium.
Postoperative complications | Up to 7 days after surgery
  Any stroke, acute renal failure (using the Kidney Disease Improving Global Outcomes (KDIGO), new-onset atrial fibrillation (more than 30 minutes or requiring cardioversion)
ICU discharge time | At ICU discharge, an average of one day after surgery
  Time and date when the patient is transferred to ward or step-down unit
Hospital discharge | At hospital discharge, an average of one week after surgery
  Time and date when the patient is discharged from the hospital
In-hospital mortality | At hospital discharge, an average of one week after surgery
  Occurrence of death during hospitalization
30-day mortality | Up to 30 days after surgery
  Occurrence of death during the first 30 days following surgery
Hospital readmission | Up to 30 days after surgery
  Need for readmission following discharge after index surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moore, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No